CLINICAL TRIAL: NCT03300583
Title: Toward a Model of Self-management; Identifying Gaps and Needs in Services for Patients With Interstitial Lung Disease
Brief Title: Toward Self-management in ILD
Status: Completed | Type: Observational
Sponsor: Kingston University (Other)
Collaborators: St. George's Hospital, London (Other); University College London Hospitals (Other)
Responsible Party: Principal Investigator, Dimitra Nikoletou, Associate Professor, Kingston University
Other Study IDs: 16.0151
Record Dates: First submitted 2017-09-28; First posted 2017-10-03 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Interstitial Lung Disease; Idiopathic Pulmonary Fibrosis; Connective Tissue Related ILD; Chronic Hypersensitivity Pneumonitis; Fibrotic Lung Disease
Keywords: Interstitial lung disease; Self-Management; Service provision
MeSH Terms: conditions — Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ILD patients: Patients from all types of ILD who are under the care of the two collaborating hospitals.
  Interventions: Behavioral: Focus groups
- Family/Carers: Family and carers of patients with ILD who are or have been treated in the two collaborating hospitals.
  Interventions: Behavioral: Focus groups
- Clinicians: Clinicians from the two collaborating hospitals and GPs from the nearby areas who treat and refer patients with ILD.
  Interventions: Behavioral: Semi-structured interviews

INTERVENTIONS:
Behavioral: Focus groups — Focus group discussion led by the PI and facilitated by another researcher.
  Groups: Family/Carers; ILD patients
Behavioral: Semi-structured interviews — 1:1 semi-structured interviews led by the PI
  Groups: Clinicians

SUMMARY:
Treating and caring for people with long term conditions accounts for a substantial proportion of health care resources. Self-management is advocated as a mechanism that can empower service users with long term conditions to choose healthier options and also transform the relationship between service user and caregivers from one in which the former is a passive recipient of care to one in which they are an active partner in decision-making.

Interstitial lung disease (ILD) is one such long term condition. Patients with ILD often express concern about the lack of information on possible rehabilitation programmes and other services that could potentially improve self-management of the disease. In addition, there is a general perception about a lack of co-ordination between health care professionals especially in relation to referral to services for comprehensive management of the disease. Therefore, the needs of patients with ILD and their carers, and possible gaps in service provision need to be explored further.

In this study, the investigators propose to explore the needs of ILD patients from all types of ILD and all stages of severity and to also involve carers and clinicians. The investigators will conduct three focus groups for patients and carers and six one-to-one interviews with clinicians to explore perceptions about service gaps and needs in two ILD centres in South and North London, UK.

This study will provide valuable information to develop the building blocks of a self-management resource and will enable the investigators to make it specific to the different types of ILD.

ELIGIBILITY:
PATIENTS

Inclusion Criteria:

* Diagnosed with Interstitial Lung disease (all types apart from sarcoidosis)
* Age >18 years
* At least one consultation with a health care professional

Exclusion Criteria:

* Diagnosed with sarcoidosis
* Unable to communicate in English
* Severity of condition and commodities preventing participation

CAREGIVERS

Inclusion Criteria:

- Currently caring for a participant with ILD

Exclusion Criteria:

- Unable to communicate in English

CLINICIANS:

Inclusion Criteria:

- Involved in the clinical management and treatment of ILD patients

Exclusion Criteria:

- Health care professionals not directly involved in management or treatment of ILD patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Interstitial Lung disease (ILD), their carers and healthcare professionals involved in their care in two hospitals in South and North London, UK.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Perceptions of service needs and gaps in current services among ILD patients, carers and clinicians | 1-2 hours
  Exploratory method, conducted using semi-structured 1:1 interviews and focus groups

SECONDARY OUTCOMES:
Differences in perceptions between participating ILD patients, carers and clinicians | 1-2 hours
  Exploratory method, conducted using semi-structured interviews and focus groups
Presentation and explanation of diagnosis and its implications to ILD patients and carers | 1-2 hours
  Exploratory method using semi-structured interviews and focus groups
Presentation and explanation of information about the management of the disease to ILD patients and carers | 1-2 hours
  Exploratory method using semi-structured interviews and focus groups
Recommended solutions for better self-management | 1-2 hours
  Exploratory method using semi-structured interviews and focus groups

CONTACTS AND LOCATIONS:
Overall Officials: Dimitra Nikoletou, PhD, Principal Investigator — Kingston University and St George's University of London- Joint Faculty- Health, Social care and Education
Locations (2):
- United Kingdom (2):
  - St George's Hospital London, London
  - University College Hospital, London

IPD SHARING:
Plan to Share IPD: No
A unique identification number will be allocated to each participant and data will not be shared without being anonymised